CLINICAL TRIAL: NCT01844310
Title: Raltegravir-based Antiretroviral Therapy for Resistant HIV-1 Infection in China
Brief Title: Raltegravir-based Antiretroviral Therapy for Resistant HIV-1 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, LI Taisheng, director of the Department of Infectious Disease, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACT1215-01
Record Dates: First submitted 2012-08-25; First posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: AIDS/HIV PROBLEM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAL +TDF+ LPV/r (Active Comparator): Arm A: RAL +TDF+ KELETRA(LPV/r) Group A will be assigned with RAL+TDF+LPV/r.
  Interventions: Drug: RAL+TDF+LPV/r
- 3TC+ TDF+LPV/r (Active Comparator): Arm B: 3TC+ TDF+KELETRA(LPV/r) Group B will be assigned with 3TC+TDF+LPV/r
  Interventions: Drug: 3TC+TDF+LPV/r

INTERVENTIONS:
Drug: RAL+TDF+LPV/r — Group A will be assigned with RAL-based regimen (RAL+TDF+LPV/r).
  Arms: RAL +TDF+ LPV/r
Drug: 3TC+TDF+LPV/r — Group B will be assigned with 3TC+TDF+LPV/r
  Arms: 3TC+ TDF+LPV/r

SUMMARY:
This study is to evaluate the safety and efficacy of RAL-based regimen in treatment-experienced patients with resistant HIV infection

DETAILED DESCRIPTION:
In our study, both efficacy and safety of raltegravir(RAL)-based therapy will be assessed. 300 treatment-experienced patients with drug-resistant HIV will be randomized to two arms (2:1). Group A (n=200) will be assigned with RAL-based regimen (RAL+TDF+LPV/r).Group B (n=100) will be assigned with current second-line regimen in China (3TC+TDF+LPV/r). Both virological and immunological profiles and responses at baseline and at week 4, 8, 12, 24, 36, and 48 will be evaluated. This study will be the first large-scale, multicenter, randomized, prospective RAL-based therapy study in China for HIV/AIDs patients. The result will provide proves for further practical antiviral therapy for China or other resource-limiting countries.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years
2. HIV seropositive and confirmed by western blot
3. have taken first line antiretroviral therapy for over one year and have any one of the criteria listed below (viral load of all the patients meeting these criteria should be confirmed at PUMCH laboratory)

   1. Viral load more than 400 copies/ml
   2. Viral rebound (confirmed by HIV RNA more than 400 copies/ml after virologic suppression)
   3. When viral load cannot be monitored, patients experience immunologic failure who meet at least one of the criteria listed below will be enrolled:

      * CD4 count equal to or lower than baseline level with first-line therapy,on two occasions over three months apart
      * CD4 count with 50 percentage fall from the on-treatment peak value
      * persistent CD4 count levels less than 100 cells/μl after over one-year antiretroviral therapy

Exclusion Criteria:

* Previous use of protease inhibitors
* Previous use of integrase inhibitors
* Pregnancy and breastfeeding
* poor compliance and drug interaction,
* opportunistic infections or malignancy at recruitment; or opportunistic infections within three months but still unstable within 14 days prior to recruitment
* HBsAg positive
* patients with the any of the following test results during screening for inclusion: WBC count<2000/μl, neutrophil count<1000/μl, Hb<9g/dl, platelet count<75000/μl, serum creatinine>1.5 ULN, transaminases or alkaline phosphatase >3 ULN, total bilirubin>2 ULN, serum creatinine kinase>2 ULN
* CCr<60 ml/min
* Current intravenous drug use
* Severe neuropathy or mental disorder
* history of alcohol abuse and unable to withdrawal
* Severe peptic ulcer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with HIV-1 RNA < 400 copies/mL at week 48 | 48 weeks

SECONDARY OUTCOMES:
Percentage of participants with HIV-1 RNA < 40 copies/mL at week 48 | 48 weeks
Change from baseline in CD4 count at week 48 | Baseline and 48 weeks
Incidence of adverse events and laboratory abnormalities in the two treatment arms from baseline to week 48 | through week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China